CLINICAL TRIAL: NCT05360108
Title: Screening for Abdominal Aortic Aneurysm and Popliteal Artery Aneurysm in At-risk Population (DAAP-PR Study)
Brief Title: Screening for Abdominal Aortic Aneurysm and Popliteal Artery Aneurysm
Acronym: DAAP-PR
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Adriano Alatri, MD, Senior Physician, Centre Hospitalier Universitaire Vaudois
Other Study IDs: DAAP-PR study
Record Dates: First submitted 2022-04-26; First posted 2022-05-04 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Aortic Aneurysm, Abdominal; Popliteal Artery Aneurysm
Keywords: Abdominal aortic aneurysm; Popliteal aneurysm; Screening
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Popliteal Artery Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational, prospective, cohort study to evaluate, by an opportunistic screening program based on vascular ultrasound, the prevalence and characteristics of Abdominal Aortic Aneurysm (AAA) and Popliteal Artery Aneurysm (PAA) in a female population as well as the prevalence and characteristics of PAA in male population.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) remains a highly topical issue given the potentially dramatic consequences associated with its rupture. In men, the prevalence of AAA is declining, probably due to improved management of risk factors. However, the most recent studies and international recommendations have reaffirmed that screening for AAA in men is still important and cost-effective. In contrast, data regarding the risk and characteristics of AAA in women are very limited and outdated. For this reason, the recommendations are contrasting and not univocal. About 35% of patients with AAA have a second aneurysm more distally. Popliteal artery aneurysm (PAA) is the most common. Like AAA, PAA is often asymptomatic and its main complication is thrombotic occlusion resulting in acute/chronic ischemia of the affected limb and a high prevalence of permanent sequelae (mainly amputation). Data on epidemiology and risk factors of PAA are very limited in men and absent in women. In addition, the benefit of PAA screening has never been assessed so far.

The aim of this study is to evaluate, by an opportunistic screening program based on vascular ultrasound, the prevalence and characteristics of AAA and PAA in a female population as well as the prevalence and characteristics of PAA in male population. The project represents the first screening program for popliteal aneurysm. Finally, the results will allow us to better assess need for and modalities of a screening program.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥65 years who are current smokers
* Men aged ≥65 years
* Women or Men aged ≥55 years with family history (first-degree relatives) for Abdominal Aortic Aneurysm (AAA) or popliteal artery aneurysm (PAA)

Exclusion Criteria:

* Patient with known diagnosis of AAA or PAA
* Patient already operated for AAA or PAA
* AAA/PAA screening or arterial assessment of lower limbs within the last 12 months
* Inability to understand and/or sign study consent
* Inability to access follow-up controls

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women or Men at high risk for aneurysmal disease
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Abdominal aortic measurement | 1 day
  Ultrasound of infrarenal aorta with diameter measured in mm
Popliteal artery measurement | 1 day
  Ultrasound of popliteal artery with diameter measured in mm

SECONDARY OUTCOMES:
Smoking habits | 1 day
  Defined by active smoking, former smoking, never smoking
Other cardiovascular risk factors | 1 day
  Arterial hypertension, Diabetes, Dyslipidemia, Obesity
History of cardiovascular diseases | 1 day
  Coronary artery disease, cerebrovascular disease, lower extremity peripheral artery disease, venous thromboembolism
Family history for aneurysmal disease | 1 day
  First-degree relatives with aneurysmal disease
Time-consuming | 1 day
  Time needed to perform screening
Surgical intervention for aneurysm | 36 months
  Number of aneurysm operated during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Mazzolai, MD, PhD, Study Chair — Centre Hospitalier Universitaire Vaudois; Adriano Alatri, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (2):
- Ospedale di Castelfranco Veneto, UOC Angiologia, Castelfranco Veneto, TV, Italy
- Centre Hospitalier Universitaire Vaudois (CHUV), Service d'Angiologie, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Chaikof EL, Dalman RL, Eskandari MK, Jackson BM, Lee WA, Mansour MA, Mastracci TM, Mell M, Murad MH, Nguyen LL, Oderich GS, Patel MS, Schermerhorn ML, Starnes BW. The Society for Vascular Surgery practice guidelines on the care of patients with an abdominal aortic aneurysm. J Vasc Surg. 2018 Jan;67(1):2-77.e2. doi: 10.1016/j.jvs.2017.10.044. PMID 29268916
- [Background] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Background] Svensjo S, Mani K, Bjorck M, Lundkvist J, Wanhainen A. Screening for abdominal aortic aneurysm in 65-year-old men remains cost-effective with contemporary epidemiology and management. Eur J Vasc Endovasc Surg. 2014 Apr;47(4):357-65. doi: 10.1016/j.ejvs.2013.12.023. Epub 2014 Jan 31. PMID 24485841
- [Background] Farber A, Angle N, Avgerinos E, Dubois L, Eslami M, Geraghty P, Haurani M, Jim J, Ketteler E, Pulli R, Siracuse JJ, Murad MH. The Society for Vascular Surgery clinical practice guidelines on popliteal artery aneurysms. J Vasc Surg. 2022 Jan;75(1S):109S-120S. doi: 10.1016/j.jvs.2021.04.040. Epub 2021 May 20. PMID 34023430
- [Background] Aboyans V, Bataille V, Bliscaux P, Ederhy S, Filliol D, Honton B, Kurtz B, Messas E, Mohty D, Brochet E, Kownator S; investigators of the E2T3A study. Effectiveness of screening for abdominal aortic aneurysm during echocardiography. Am J Cardiol. 2014 Oct 1;114(7):1100-4. doi: 10.1016/j.amjcard.2014.07.024. Epub 2014 Jul 18. PMID 25127549
- [Background] Matsumura Y, Ochi Y, Wada M, Hirakawa D, Yamanaka S, Kamioka M, Kitaoka H, Orihashi K, Nakaoka Y, Doi Y, Sugiura T. Usefulness of Screening for Abdominal Aortic Aneurysm During Transthoracic Echocardiography in Women >/=50 Years of Age. Am J Cardiol. 2018 Dec 15;122(12):2147-2150. doi: 10.1016/j.amjcard.2018.08.050. Epub 2018 Sep 22. PMID 30360889